CLINICAL TRIAL: NCT02396407
Title: Spillover Effects of Water, Sanitation, and Hygiene Interventions on Child Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other); Stanford University (Other); Bill and Melinda Gates Foundation (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1R21HD076216-01A1 (NIH); 1R21HD076216-01A1 (NIH)
Record Dates: First submitted 2015-03-18; First posted 2015-03-24 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Helminthiasis; Diarrhea; Respiratory Infection
Keywords: Chlorine water treatment; Point-of-use water treatment; Household water treatment with safe storage; Handwashing with soap; Hand hygiene; Latrines; Child potties; Intestinal parasitic infection; Soil-transmitted helminths; Water; Sanitation; Handwashing; Diarrhea; Herd immunity; Helminths
MeSH Terms: conditions — Helminthiasis; Diarrhea; Respiratory Tract Infections; Intestinal Diseases, Parasitic | interventions — Sanitation; Hygiene

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Combined water, sanitation, and hygiene (Active Comparator): Water quality, Sanitation, Handwashing
  Interventions: Behavioral: Combined water, sanitation, and hygiene
- Non-intervention arm (No Intervention): None. Households will continue their usual practices.

INTERVENTIONS:
Behavioral: Combined water, sanitation, and hygiene — Water: Free chlorine tablets (Aquatabs; NaDCC) and safe storage vessel to treat and store drinking water.
  Sanitation: Free child potties, sani-scoop hoes to remove feces from household, and latrine upgrades to a dual pit latrine for all households in study compounds.
  Handwashing: Handwashing stations including soapy water bottles and detergent soap.
  Local promoters visit study compounds at least monthly to deliver behavior change messages that focus on (1) treating drinking water for children < 36 months of age, (2) use of latrines for defecation and the removal of human and animal feces from the compound, and (3) handwashing with soap at critical times around food preparation, defecation, and contact with feces.
  Arms: Combined water, sanitation, and hygiene

SUMMARY:
The purpose of this study is to measure whether a combined water, sanitation, and hygiene intervention leads to improved health of children who did not receive the intervention themselves and who live within a close vicinity of intervention recipients.

DETAILED DESCRIPTION:
Almost 90% of diarrhea cases and 15% of under-5 diarrhea deaths worldwide could be prevented through improved water, sanitation, and hygiene. Sanitation interventions are also important for the prevention of soil-transmitted helminths, which infect 21 million children under five each year. Infection with soil-transmitted helminths and repeated episodes of diarrhea early in life can compromise physical and cognitive growth and development, resulting in poorer school performance later in life. Thus, water, sanitation, and hygiene (WASH) interventions are important not only for reducing child mortality, but also for preventing cycles of poverty and poor health.

It is possible that WASH interventions affect not only those who receive them but also those who are geographically proximate or connected socially to those receiving the intervention. Indeed, there is a large infectious disease modeling literature based on this premise. Investigators define intervention effects on non-recipients "spillovers", and they are often referred to as "herd effects" or "indirect effects". Most studies that have empirically measured spillovers of child health interventions with an experimental design have focused on vaccines and deworming, and no studies have measured spillovers from WASH interventions. The development and application of methodology for measuring spillovers of community interventions empirically would make a valuable contribution to fields including epidemiology, economics, political science, and social welfare, all of which are concerned with measuring the impact of programs and interventions which may spill over. The presence and magnitude of positive spillovers are important; if spillovers are present and are in the same direction as treatment effects but are not accounted for when estimating treatment effects, estimates will be biased towards the null. As a result, both the efficacy and cost effectiveness of the intervention will be underestimated.

In this study, investigators will measure spillovers of water, sanitation, and hygiene interventions in an existing, large, rigorously designed trial: the WASH Benefits trial (https://clinicaltrials.gov/ct2/show/NCT01590095). Funded by the Bill & Melinda Gates Foundation, this trial aims to measure the individual and combined effects of water, sanitation, and hygiene interventions on child health and development. It is a cluster-randomized, controlled trial with six treatment arms and a double-sized control arm carried out in rural Bangladesh. This add-on study is funded by the National Institute for Child Health and Human Development (1R21HD076216-01A1). Investigators hypothesize that children who live in close proximity to compounds that receive a combined sanitation, handwashing, and water treatment intervention--compared to children who live in close proximity to control compounds (no intervention)--will have: 1) lower prevalence of diarrhea, 2) lower prevalence and intensity of infection of soil transmitted helminths, and 3) lower prevalence of respiratory illness.

Investigators will collect additional data from the existing combined intervention (sanitation+handwashing+water) and control arms of the WASH Benefits trial. For each WASH Benefits household, investigators will locate the nearest household with children 0-59 months of age that are not enrolled in WASH Benefits and collect data in that household. Our primary outcomes are soil transmitted helminth infection among children 0-59 months, caregiver-reported 7-day diarrhea, and respiratory illness among children 0-59 months (the same age as the WASH Benefits cohort). Our findings will document either the presence or absence of spillovers of the combined sanitation+handwashing+water intervention.

ELIGIBILITY:
Inclusion Criteria:

* Children not enrolled in WASH Benefits who live in a compound within 120 steps (2 minutes walking time) of a compound enrolled in WASH Benefits (combined WSH or control arms) and are 0-60 months 24 months after intervention

Exclusion Criteria:

* Children enrolled in WASH Benefits
* Children who live in compounds (baris) that share a courtyard with a compound enrolled in the WASH Benefits study
* Children who live in compounds (baris) that share a latrine or handwashing station with a compound enrolled in the WASH Benefits study

Max Age: 60 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1789 (Actual)
Dates: Start 2015-01; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Prevalence of soil-transmitted helminths (Ascaris, hookworm, Trichuris) | Measured approximately 24 months after intervention
  Children's stool will be collected. Kato-Katz will be used to detect Ascaris, hookworm, Trichuris ova in stool. Stool samples with any ova will be considered positive.
Intensity of soil-transmitted helminth infections (Ascaris, hookworm, Trichuris) | Measured approximately 24 months after intervention
  Children's stool will be collected. Kato-Katz will be used to detect Ascaris, hookworm, Trichuris ova in stool. Intensity will be measured using WHO cutoffs based on the number of eggs per gram of stool (>=5,000 eggs/gram for Ascaris, >=1,000 eggs/gram for hookworm, and >=2,000 eggs/gram for Trichuris).

SECONDARY OUTCOMES:
Diarrhea prevalence | Measured approximately 24 months after intervention
  Diarrhea is defined as 3+ loose or watery stools in 24 hours or 1+ stools with blood in 24 hours. Diarrhea will be measured in interviews using caregiver-reported symptoms with 2-day and 7-day recall, measured 24 months after intervention.
Respiratory illness prevalence | Measured approximately 24 months after intervention
  Respiratory illness is defined as a persistent cough or difficulty breathing in the 7 days before the interview. Respiratory illness will be measured in interviews using caregiver-reported symptoms with 2-day and 7-day recall, measured 24 months after intervention.

CONTACTS AND LOCATIONS:
Overall Officials: John M Colford, Jr., MD PhD, Principal Investigator — University of California, Berkeley
Locations (1):
- International Centre for Diarrhoeal Disease Research, Bangladesh, Dhaka, Bangladesh

REFERENCES:
- [Background] Arnold BF, Null C, Luby SP, Unicomb L, Stewart CP, Dewey KG, Ahmed T, Ashraf S, Christensen G, Clasen T, Dentz HN, Fernald LC, Haque R, Hubbard AE, Kariger P, Leontsini E, Lin A, Njenga SM, Pickering AJ, Ram PK, Tofail F, Winch PJ, Colford JM Jr. Cluster-randomised controlled trials of individual and combined water, sanitation, hygiene and nutritional interventions in rural Bangladesh and Kenya: the WASH Benefits study design and rationale. BMJ Open. 2013 Aug 30;3(8):e003476. doi: 10.1136/bmjopen-2013-003476. PMID 23996605
- [Background] Lin A, Arnold BF, Afreen S, Goto R, Huda TMN, Haque R, Raqib R, Unicomb L, Ahmed T, Colford JM, Luby SP. Household environmental conditions are associated with enteropathy and impaired growth in rural Bangladesh. Am J Trop Med Hyg. 2013 Jul;89(1):130-137. doi: 10.4269/ajtmh.12-0629. Epub 2013 Apr 29. PMID 23629931
- [Background] Sultana R, Mondal UK, Rimi NA, Unicomb L, Winch PJ, Nahar N, Luby SP. An improved tool for household faeces management in rural Bangladeshi communities. Trop Med Int Health. 2013 Jul;18(7):854-60. doi: 10.1111/tmi.12103. Epub 2013 Apr 5. PMID 23557125
- [Background] Hulland KR, Leontsini E, Dreibelbis R, Unicomb L, Afroz A, Dutta NC, Nizame FA, Luby SP, Ram PK, Winch PJ. Designing a handwashing station for infrastructure-restricted communities in Bangladesh using the integrated behavioural model for water, sanitation and hygiene interventions (IBM-WASH). BMC Public Health. 2013 Sep 23;13:877. doi: 10.1186/1471-2458-13-877. PMID 24060247
- [Background] Dreibelbis R, Winch PJ, Leontsini E, Hulland KR, Ram PK, Unicomb L, Luby SP. The Integrated Behavioural Model for Water, Sanitation, and Hygiene: a systematic review of behavioural models and a framework for designing and evaluating behaviour change interventions in infrastructure-restricted settings. BMC Public Health. 2013 Oct 26;13:1015. doi: 10.1186/1471-2458-13-1015. PMID 24160869
- [Background] Vujcic J, Ram PK, Hussain F, Unicomb L, Gope PS, Abedin J, Mahmud ZH, Islam MS, Luby SP. Toys and toilets: cross-sectional study using children's toys to evaluate environmental faecal contamination in rural Bangladeshi households with different sanitation facilities and practices. Trop Med Int Health. 2014 May;19(5):528-36. doi: 10.1111/tmi.12292. Epub 2014 Mar 19. PMID 24645919
- [Background] Ercumen A, Naser AM, Unicomb L, Arnold BF, Colford JM Jr, Luby SP. Effects of source- versus household contamination of tubewell water on child diarrhea in rural Bangladesh: a randomized controlled trial. PLoS One. 2015 Mar 27;10(3):e0121907. doi: 10.1371/journal.pone.0121907. eCollection 2015. PMID 25816342
- See also: WASH Benefits Bangladesh ClinicalTrials.gov Registration — https://clinicaltrials.gov/ct2/show/NCT01590095
- See also: Description of the design and rationale for WASH Benefits (open access article) — http://bmjopen.bmj.com/content/3/8/e003476.full